CLINICAL TRIAL: NCT04772560
Title: Toric Contact Lens Digital Performance and Comfort Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kathryn Richdale (Other)
Responsible Party: Sponsor-Investigator, Kathryn Richdale, Associate professor, University of Houston
Organization: University of Houston (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00002753
Record Dates: First submitted 2021-02-23; First posted 2021-02-26 (Actual); Results first posted 2022-03-10 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-02

CONDITIONS: Astigmatism
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Toric, Then Sphere (Experimental): Participants who received Toric contact lenses first and spherical lenses after 10 days
  Interventions: Device: Precision1 for Astigmatism; Device: Precision1 Sphere
- Sphere, Then Toric (Experimental): Participants who received Spherical contact lenses first and Toric lenses after 10 days
  Interventions: Device: Precision1 for Astigmatism; Device: Precision1 Sphere

INTERVENTIONS:
Device: Precision1 for Astigmatism — Daily disposable soft toric contact lens
Device: Precision1 Sphere — Daily disposable soft spherical contact lens

SUMMARY:
This study seeks to quantify digital visual performance and subjective visual acceptance of toric contact lenses as compared to spherical lenses in low to moderate astigmatic patients.

DETAILED DESCRIPTION:
This study seeks to quantify the near visual performance and subjective visual acceptance of toric contact lenses as compared to spherical lenses in an astigmatic cohort of patients. Primary Hypotheses: Subjects will have better near visual acuity and near visual performance with toric, as opposed to spherical, contact lens correction. As such, the following hypotheses will be tested: H01: There is no statistically significant difference in near visual acuity or near vision performance between contact lenses corrections Ha1: There is a statistically significant difference in visual acuity or vision performance between contact lenses corrections

ELIGIBILITY:
Inclusion Criteria:

* 18 to 39 years of age (inclusive)
* pl to -6.00D vertexed sphere power and -0.75 to -1.50D vertexed refractive cylinder OD and OS
* Current/established full time (>6 days week, >8 hours/day) soft contact lens wearer
* Best corrected acuity of 20/25 or better in each eye
* Self-report of at least 4 hrs/day using digital devices
* Willing to wear lenses at least 8 hours each day during the study period
* Able to speak and read English at a high school level / have at least a high school diploma or equivalent (by self-report)

Enclusion Criteria:

* History of ocular pathology or surgery
* Binocular vision disorder (i.e., tropia, convergence or accommodative insufficiency)
* Gas permeable lens wear for at least 3 months
* Symptomatic soft contact lens wearer (CLDEQ-8 score <12 at baseline)

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-03-16 (Actual); Primary Completion 2021-12-13 (Actual); Study Completion 2021-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Richdale, Principal Investigator — University of Houston College of Optometry
Locations (1):
- University of Houston College of Optometry, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 30 participants were screened for eligibility between March and December 2021
Pre-assignment Details: 23 of 30 participants were randomized. Of those not randomized, 7 did not meet inclusion criteria.
Groups:
- Toric Then Spherical: Participants who received toric contact lenses first and spherical lenses after 10 days
- Spherical Then Toric: Participants who received spherical contact lenses first and toric lenses after 10 days
Period: Overall Study
Arm/Group | Toric Then Spherical | Spherical Then Toric
Started | 11 | 12
Completed | 11 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 7 participants were screen failed.
Groups:
- All Participants: 23 participants who had completed the study
Arm/Group | All Participants
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.4 (4.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 8
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Near Visual LogMAR Acuity
Description: High contrast LogMAR visual acuity was assessed at 40 cm using the M&S Clinical Trial Suite system (Niles, Illinois, USA). The system was calibrated according to the manufacturer's directions every day, prior to use. Testing was performed binocularly 10+/-2 days after each intervention. The test started at 20/60 and continued until three letters were missed on a line.
Time Frame: 10 +/- 2 days
Measure: Mean (Standard Error); unit: LogMAR
Arm/Group | All Participants
Number analyzed (Participants) | 23
LogMAR
  Toric CL | -0.10 (0.02)
  Spherical CL | -0.03 (0.21)

2. Primary Outcome: Dynamic Visual Acuity
Description: Dynamic VA was determined using a custom-made iPad application. The subject was instructed to hold the iPad at 40cm and presented with a Landolt C surrounded by crowding bars for 0.3s each, starting from 0.5 LogMAR and progressing to smaller sizes using a staircase threshold method. Testing was performed binocularly 10+/-2 days after each intervention
Time Frame: 10 +/- 2 days
Measure: Mean (Standard Error); unit: LogMAR
Arm/Group | All Participants
Number analyzed (Participants) | 23
LogMAR
  Toric CL | 0.04 (0.02)
  Spherical CL | 0.11 (0.02)

ADVERSE EVENTS:
Time Frame: 10 ± 2 days for each intervention
Description: AE information was collected at each study visit
Groups:
- Toric Contact Lens Wear; Spherical Contact Lens Wear: 23 participants had completed the study
Arm/Group | Toric Contact Lens Wear | Spherical Contact Lens Wear
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 4/23 | 0/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Toric Contact Lens Wear (N=23) | Spherical Contact Lens Wear (N=23)
Corneal staining (Eye disorders) | 3 (3) | 0 (0) — Corneal staining > Grade 2 (CCLRU scale)
Hordeolum (Eye disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2021-08-18): https://cdn.clinicaltrials.gov/large-docs/60/NCT04772560/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2021-12-20): https://cdn.clinicaltrials.gov/large-docs/60/NCT04772560/SAP_001.pdf